CLINICAL TRIAL: NCT00041704
Title: A Phase 2 Open-Label Study of the Safety and Efficacy of Intravenous Anidulafungin as a Treatment for Azole-Refractory Mucosal Candidiasis.
Brief Title: The Safety and Efficacy of Intravenous Anidulafungin as a Treatment for Azole-Refractory Mucosal Candidiasis (FRMC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Vicuron Pharmaceuticals (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VER002-11; A8851004
Record Dates: First submitted 2002-07-12; First posted 2002-07-16 (Estimated); Last update posted 2008-10-20 (Estimated); Status verified 2008-10

CONDITIONS: Candidiasis
Keywords: Azole-Refractory Mucosal Candidiasis; Mucosal Candidiasis
MeSH Terms: conditions — Candidiasis | interventions — Anidulafungin

INTERVENTIONS:
Drug: Anidulafungin, VER002

SUMMARY:
Anidulafungin is an antifungal agent of the echinocandin class which is highly active in vitro against fluconazole resistant Candida species. The efficacy of anidulafungin has demonstrated in various animal models of fluconazole-resistant mucosal disease; as well as, in Phase 2 Esophageal Candidiasis studies. This study is intended to offer patients with FRMC an alternate therapy with amphotericin B or with other agents whose efficacy and/or safety are inadequate in the treatment of this disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of definite azole-refractory mucosal candidiasis (oral or oropharyngeal candidiasis or esophageal candidiasis), i.e., patients who have not responded to a prior 14-day course of fluconazole at a dose of at least 200 mg daily or other azole (e.g. voriconazole)
* Grade 1 or higher mucosal disease and microscopic or culture confirmation of yeast

Exclusion Criteria:

* Pregnant female
* Hypersensitivity to anidulafungin or echinocandin therapy
* Hypersensitivity to Tween 80 (polysorbate 80) or tartaric acid
* Abnormal blood chemistries: Bilirubin >2 times the upper limit of normal; AST (aspartate aminotransferase) or ALT (alanine aminotransferase) > 4 times the upper limit of normal
* Less than four weeks since prior participation in an investigational drug or device study with the exception of antiretroviral agents or licensed agents
* Patients taking other systemic antifungal therapies while on this study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2002-08; Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Versicor, Inc., King of Prussia, Pennsylvania, United States